CLINICAL TRIAL: NCT02514707
Title: Outcomes of HIV Infected Individuals After Ten Years on Antiretroviral Treatment
Acronym: ART Long Term
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Infectious Diseases Institute (Other)
Responsible Party: Sponsor-Investigator, Infectious Diseases Institute, Principal Investigator, Makerere University
Organization: Makerere University (Other)
Other Study IDs: ST/0113/15
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma (4 aliquots), serum (4 aliquots), packed cells pellets (5 aliquots) for each patient
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Title: Outcomes of HIV infected individuals after ten years on antiretroviral treatment Short Title/Study ID: ALT cohort Protocol Version and Date: Version 1.0 June 2013 Clinical Phase: NA Methodology: Prospective observational study Study Duration: 01 January 2014- 30th June 2025 Study Centre(s): Single centre (Infectious Diseases Institute, Kampala, Uganda) Number of Subjects: Enrollment of 1,000 study participants. All patients discharged from the IDI Research cohort (10 years of follow up on ART) will be offered to participate in the study. Additional patients with similar characteristics will be enrolled from he clinic Diagnosis and Main Inclusion Criteria: HIV patients above 18 years and in their 10th year of ART Main Exclusion Criteria: ART started outside IDI Study Product, Dose, Route, Regimen: ART will be provided according to standard of care at IDI and according to the WHO and Ugandan guidelines Duration of follow up: 10 years Reference therapy, Dose, Route, Regimen: Not applicable Recruitment Schedule: 1 January 2014- 30 June 2015 Statistical Methodology: Time to event analysis (end of treatment, failure, death, switch, occurrence of drug toxicities) including Kaplan-Meier curves and Cox regression will be performed. Endpoints will be correlated with characteristics at ART start and at study enrollment. Possible confounding variables, if available, will be considered.

GCP Statement: This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, and ICH-GCP as well as all national legal and regulatory requirements.

DETAILED DESCRIPTION:
1. INTRODUCTION: 1.1. Disease Setting/Patient Population: Advances in HIV antiretroviral therapy (ART) have dramatically reduced mortality from HIV, primarily because of the reduction in deaths attributable to AIDS defining conditions such that a person receiving state-of-the-art ART may now expect to live 25 years and potentially longer. However the number of deaths attributable to causes not conventionally considered to be HIV related is increasing with up to 50% of all patients with HIV die from causes considered unrelated to HIV. Thus, management of HIV now involves the treatment of chronic diseases with the possibility of near normal life expectancy, but often with multiple co morbidities.

1.2. Background and Rationale: Cardiovascular risk in patients on ART Metabolic complications, including dyslipidemia, insulin resistance, and altered fat distribution (loss of subcutaneous fat and a relative increase in central fat), are common in adults infected with HIV who are receiving ART. These complications may increase these patients' risk of cardiovascular disease. Recent studies suggest that some types of ART may be associated with increased risk of cardiovascular disease, a cause for concern given that people living with HIV may take ART for decades. The mechanisms causing an increased risk of cardiovascular disease are unclear, but it has been suggested that it may relate to dyslipidemia, insulin resistance, diabetes mellitus, inflammation, impaired fibrinolysis, factors specific to antiretroviral medications, or combinations of these factors. Grinspoon and Carr further speculate that both HIV and ART might be associated with many of these risk factors.

From observational data the evidence linking ART and cardiovascular disease has pointed specifically to PIs as a class since they may promote the formation of atherosclerotic lesions, and other NRTI specific agents (abacavir, didanosine). However up to date the role of abacavir remain controversial. All potential cardiovascular risk factors, including dyslipidemia, insulin resistance, hypertension, smoking, sedentary lifestyle, weight, and family history, should be assessed. Ideally glucose levels and fasting lipid levels should be checked annually in all HIV patients on ART.

Renal disease The use of combination, highly active antiretroviral therapy (HAART) since the mid-1990s has resulted in significant and sustained reductions in morbidity and mortality from HIV infection, including significant declines in HIV-associated nephropathy (HIVAN). At the same time, however, a variety of ART-related renal side effects have been noted, including proteinuria and renal tubular damage, interstitial nephritis, nephrolithiasis, and overall declines in glomerular filtration rate. Kidney function has been estimated to be abnormal in up to 30% of HIV-infected patients. In addition, other metabolic complications such as type 2 diabetes and hypertension may also contribute to renal dysfunction over time.

In Sub- Saharan Africa, including Uganda, tenofovir has been included as one of the recommended drugs for first line regimens, due to its comparable efficacy to other first-line regimens containing stavudine, zidovudine or abacavir, and has the additional advantage of low toxicity and availability as a once-daily, fixed-dose generic formulation. Yet concerns regarding its renal tubular toxicity remain especially on its use in resource-limited settings where clinical detection of renal impairment is difficult in. Early stages of renal dysfunction can be are assessed through laboratory monitoring of creatinine and glomerular filtration rate. Current guidelines contraindicate TDF use when creatinine clearance (CrCl) falls below 50 ml/min unless dose reductions are made. If TDF is to be implemented in resource-limited settings where numbers requiring antiretroviral therapy are high but access to laboratory services are scarce, these monitoring protocols may need to be further simplified. Ideally in order to monitor patients for renal toxicity, It is recommended that urinalysis for proteinuria is performed routinely and creatinine clearance calculated; co morbidities that may contribute to elevated risk of kidney disease should be also closely monitored. Data from the DART trial, a prospective randomized clinical trial conducted in an African setting, showed a low (1.3%) rate of severe renal impairment through 96 weeks, with no difference in TDF-containing and non TDF-containing regimens. Similarly data from a routine program setting (Lesotho) shows that renal toxicity due to tenofovir is rare and mild.

Late mortality:

A multicenter cohort study from Europe and North America reported that already after 4 years on ART the cumulative incidence of non-AIDS-related deaths exceeded that of AIDS-related deaths. The most frequent non-AIDS causes of death were non-AIDS malignancy (11.8%), non-AIDS infection (8.2%), cardiovascular disease (7.9%, of which 40% were myocardial infarction/ischemic heart disease and 18% stroke), violence (7.8%, including suicide, substance abuse, and homicide/accident/unspecified), and liver disease (7.1%, of which 55.8% were hepatitis related). The most frequent sites for non-AIDS malignancies were respiratory tract or intrathoracic organs (36.7%); digestive organs and peritoneum (28.7%); lip, oral cavity, and pharynx (6.0%); and skin (4.7%).

Rationale for this study:

Little information is available on patients on ART for a long term period from Sub-Saharan Africa. Particularly no information is available on long term complications of ART and non HIV related events. Although data is available from resource rich settings, this information may not be applicable to Sub-Saharan Africa due to the different antiretroviral treatment drugs used and ART monitoring strategies, different HIV subtypes, as well as different ethnicity and endemic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
3. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
4. On the 10th consecutive year on ART (any combination including second line)

Exclusion Criteria:

1. ART started before registration in the IDI clinic
2. Subjects enrolled in an experimental clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on ART for more than 9 years receiving care and treatment through the adult clinic at the Infectious Diseases Institute in Kampala, Uganda
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the clinical profile of patients (CD4 cell count, viral loads, WHO state, history of OIs, previous use of ART, level of anemia, and other medical conditions, drug mutations) | Baseline
  A cross sectional analysis at study enrollment will be performed to characterize the clinical profile of patients after at least 9 years on ART including CD4 cell count, viral loads, WHO state, history of OIs, previous use of ART, level of anemia, and other medical conditions, drug mutations.
Drug toxicity as any grade 3 & 4 DAD Scale | Yearly for 10years
  To determine the incidence of side effects and drug toxicity, requirement for drug switches, development of opportunistic infections (OIs) (in particular tuberculosis), morbidity (particularly non HIV related morbidity such as cancer and cardiovascular diseases), medication adherence and loss to follow up; to determine the relationship between various clinical and demographic variables at initiation of treatment and cohort enrollment and subsequent outcome.
Causes of mortality | Yearly for 10years
  To investigate causes of mortality using a standardized collection tool for verbal autopsies

SECONDARY OUTCOMES:
Composite measure of change in Sexual Behavior over time | Yearly for 10years
  To assess sexual behavior and sexual networks by routinely administered questionnaires through nurse counselors as well as to document over time the sero-status of the partners.
Variation of drug levels due to drug-drug interaction | Yearly for 10years
  To investigate drug-drug interactions between antiretroviral drugs and concomitant medicines that are used by a sub-group of cohort subjects
Cost Analysis | Yearly for 10years
  To investigate cost (cost analysis) of care of patients on long term ART and compare it with the cost of care of patients on short and middle (<10 years) ART.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Castelnuovo, MD, PhD, Study Director — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute, Kampala, Kampala, Uganda